CLINICAL TRIAL: NCT04757597
Title: Safety and Efficacy of Remote Ischemic Conditioning in Patients With Cerebral Amyloid Angiopathy-related Intracerebral Hemorrhage:A Multicenter, Randomized, Controlled Study
Brief Title: Remote Ischemic Conditioning for Cerebral Amyloid Angiopathy-related Intracerebral Hemorrhage
Acronym: RIC-CAAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Collaborators: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other); Bejing Fengtai You'anmen Hospital (Unknown)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIC-CAAH
Record Dates: First submitted 2021-02-13; First posted 2021-02-17 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Intracerebral Hemorrhage Lobar; Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): RIC treatment and regular treatment.
  Interventions: Device: Remote ischemic conditioning
- Regular treatment (No Intervention): Regular treatment alone.

INTERVENTIONS:
Device: Remote ischemic conditioning — RIC is a non-invasive therapy that performed by an electric autocontrol device with cuff placed on arm. RIC procedures consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on one arm. The procedure will be performed once daily for consecutive 10-14 days after enrollment.
  Arms: RIC group

SUMMARY:
Cerebral amyloid angiopathy-related intracerebral (CAAH) hemorrhage is second factor of primary intracerebral hemorrhage. However, no effective prevention and treatment strategies have been established. Remote ischemic conditioning is a neuroprotective strategy. In animal studies，RIC is efficiency in accelerating the absorption of hematoma. Therefore, the investigators plan to carry out this research to evaluate the safety and efficacy of RIC in patients with CAA related ICH.

DETAILED DESCRIPTION:
In China, primary intracerebral hemorrhage accounts for 80-85% of all types of intracerebral hemorrhage, while cerebral amyloid angiopathy-related intracerebral hemorrhage is the second factor, accounting for approximately 20-30%. It is often characterized by repeated and multifocal lobar hemorrhage, which will not only cause neurological deficit on the limbs, but also influence the cognitive level of patients and may even be life-threatening. At present, the role of surgery in CAA-related ICH is controversial, and there is no effective prevention and treatment strategies have been established. Additionally, it is always associated with a low rate of good prognosis(11%-60%) and a high risk of recurrent ICH (10%-60%). Thus, a novel approach which can improve the clinical outcome and reduce the risk of recurrent intracerebral hemorrhage is urgently needed.

Remote ischemic conditioning (RIC) has been developed as a neuroprotective strategy to prevent and treat acute ischemic stroke and small cerebrovascular disease. Additionally, clinical research testified that RIC is safe and feasible for patients with subarachnoid hemorrhage. In animal studies, RIC is efficiency in accelerating the absorption of hematoma. Therefore, the investigators plan to carry out this research to evaluate the safety and efficacy of RIC in patients with CAA related ICH.

ELIGIBILITY:
Inclusion Criteria:

* Age≥55 and ≤85.
* The diagnosis of single or multiple spontaneous lobar cerebral hemorrhage is confirmed by brain CT scan(defined as possible or probable CAA by the Boston criteria) .
* Hematoma volume of 10 to 50 ml.
* Glasgow Coma Score (GCS)>8.
* Without surgery.
* Starting RIC treatment between 24 and 48 hours of ictus.
* Signed and dated informed consented is obtained.

Exclusion Criteria:

* Patients with suspected secondary ICH related to tumor, coagulopathy, ruptured aneurysm or arteriovenous malformation, or venous sinus thrombosis.
* ICH concomitant with intraventricular hemorrhage, subdural hematoma, epidural hematoma subarachnoid hemorrhage or the condition of unstable vital signs which may be life-threatening.
* Evidence of significant shift of midline brain structure (>5mm) or herniation on brain imaging.
* Contraindication to MRI scan, such as intracranial metal implants, cardiac pacemaker, severe claustrophobia, history of seizures and so on
* Patients with a pre-existing neurological deficits (modified Ranks scale score >2) or psychiatric disease that would confound the neurological or functional evaluations.
* Use of warfarin or heparin within 7 days before the baseline visit
* Contraindication for remote ischemic conditioning: severe soft tissue injury, limb deformities, fracture, atrial fibrillation or peripheral vascular disease in the upper limbs.
* Life expectancy of less than 1 year due to co-morbid conditions.
* Severe, sustained hypertension (SBP > 180 mmHg or DBP > 110 mmHg).
* Severe hepatic and renal dysfunction.
* Known pregnancy (or positive pregnancy test), or breast-feeding.
* Concurrent participation in another research protocol for investigation of another experimental therapy.
* Any condition which, in the judgment of the investigator, might increase the risk to the patient.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 90±7 days
  Safety

SECONDARY OUTCOMES:
Changes of intracerebral hematoma volume | 14± 2 days
  Intracerebral hematoma volume (ml) is assessed by CT brain scan.
Changes of perihematomal edema volume | 14± 2 days
  Perihematomal edema volume (ml) is assessed by CT brain scan.
Incidence rate of the perihematomal edema expansion | 14± 2 days
  The enlargement of perihematomal edema volume (ml) is assessed by CT brain scan.
Shift of midline brain structure | 14± 2 days
  Shift of midline brain structure (mm) is assessed by CT brain scan
Prognosis of function outcome at 90 Days | 90±7 days
  accessed by modified Rankin score
Prognosis of neurological function at 90 Days | 90±7 days
  The Barthel index will be assessed at follow-up.
Changes of serum biomarker of blood brain barrier (Matrix metalloproteinases，MMPs) | 7± 2 days
  The biomarker of blood brain barrier（MMPs） are assemented by the same laboratory.
Changes of serum biomarker of inflammatory ( interleukin) | 7± 2 days
  The interleukin will be assemented by the same laboratory.
Other adverse events related to RIC treatment | 90±7 days
  Other adverse events related to RIC treatment,such as mucocutaneous hemorrhage,changes in coagulation function and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamada M. Cerebral amyloid angiopathy: emerging concepts. J Stroke. 2015 Jan;17(1):17-30. doi: 10.5853/jos.2015.17.1.17. Epub 2015 Jan 30. PMID 25692104
- [Background] Arima H, Tzourio C, Anderson C, Woodward M, Bousser MG, MacMahon S, Neal B, Chalmers J; PROGRESS Collaborative Group. Effects of perindopril-based lowering of blood pressure on intracerebral hemorrhage related to amyloid angiopathy: the PROGRESS trial. Stroke. 2010 Feb;41(2):394-6. doi: 10.1161/STROKEAHA.109.563932. Epub 2009 Dec 31. PMID 20044530